CLINICAL TRIAL: NCT06196177
Title: Regulation of Cardiac Function After TAVR in Patients With Severe Aortic Stenosis Combined With Cardiac Insufficiency: a Prospective, Single-center, Randomized Controlled Study
Brief Title: Effects of Levosimendan on Cardiac Function After TAVR in Patients With Heart Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202309-008
Record Dates: First submitted 2023-12-13; First posted 2024-01-09 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Aortic Stenosis, Severe
MeSH Terms: conditions — Heart Failure; Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levosimontane group (Experimental): name：Levosimendan injection dose：12.5mg；once；24h
  Interventions: Drug: Levosimontane injection
- control group (No Intervention): blank control

INTERVENTIONS:
Drug: Levosimontane injection — Levosimendan injection was given once intravenously with a micro-pump: 12.5mg levosimendan injection was diluted with 5% glucose injection to 50ml at the initial pump speed of 2ml/h for 24h.
  Other Names: wen，yue
  Arms: Levosimontane group

SUMMARY:
Patients with severe aortic stenosis combined with severe heart failure often miss the opportunity for surgery, and the prognosis is poor with drug therapy alone.In recent years, the emergence of transcatheter aortic valve replacement (TAVR) has brought new hope for these patients, and since its birth in 2002, TAVR has been widely used internationally, and its safety and efficacy have been confirmed by several large, prospective, randomized controlled studies.

Levosimendan is a new type of positive inotropic drug. It not only enhances myocardial contractile force through calcium sensitization, but also activates K+ sensitive channel KATP on the membrane of vascular smooth muscle, relaxes the arteries and veins of the whole body, and reduces the front and back load of the heart, pulmonary vascular resistance and systemic vascular resistance. A series of studies suggested that for patients undergoing thoracotomy in various cardiac surgeries, regardless of whether the patients were accompanied by ventricular systolic dysfunction before surgery, the use of levosimendan resulted in significantly higher postoperative cardiac function and decreased mortality than the control group, and patients with preoperative LVEF < 40% benefited more.

At present, there are no studies to clarify the regulatory effect of levosimendan on cardiac function after TAVR in patients with severe aortic stenosis complicated with cardiac insufficiency. This is a randomized controlled study. On the basis of basic drug therapy, the treatment group was given levosimendan to analyze the regulatory effect of levosimendan on cardiac function after TAVR.

DETAILED DESCRIPTION:
We plan to recruit 112 patients with severe aortic stenosis and cardiac insufficiency, which，after TAVR, were randomly divided into treatment group (56 cases, intravenous levosimendan) and control group (56 cases).

The treatment group was given levosimendan injection intravenously once: 12.5mg levosimendan injection was diluted to 50ml with 5% glucose injection, the initial pump speed was 2ml/h, and maintained for 24 hours.

In the process of drug q1h monitoring blood pressure. If the systolic blood pressure was lower than 90mmHg, the blood pressure was remeasured 5 minutes later. If the systolic blood pressure was still lower than 90mmHg, 10mg norepinephrine injection +45ml 5% glucose injection was given intravenously by micro pump, the initial 2ml/h. The blood pressure was monitored, and the pump speed was adjusted according to the blood pressure to maintain the systolic blood pressure at 90-110mmHg.

Preoperative and postoperative immediately, after 3 days and postoperative 1 month, electrocardiogram, echocardiography and venous blood. Three tubes of venous blood were collected each time, and each tube was sent to the laboratory department of Qilu Hospital for blood routine, liver and kidney function, blood biochemistry, NT-proBNP and troponin I detection. The remaining samples were destroyed immediately after detection. The results of 6-minute walk test and the incidence of cardiovascular events were recorded at 1 month after operation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 65-85 years undergoing TAVR;
* Echocardiography diagnosed severe aortic valve stenosis with LVEF<0.4；
* Prior to the initiation of the study, the patients or their legal representatives signed the informed consent form.

Exclusion Criteria:

* Adverse reactions to levosimendan or other excipients;
* In addition to the aortic valve disease, still with cardiac mechanical obstructive diseases;
* Patients with severe hepatic and renal impairment (creatinine clearance <30ml/min);
* Patients with severe hypotension (SBP<90mmHg or DBP<60mmHg) and ventricular tachycardia, ventricular fibrillation, and frequent premature ventricular contractions.
* Severe complications occurred during TAVR.
* Are involved in other clinical studies
* Other clinically significant respiratory, digestive, hematological, infectious, immune, endocrine, neuropsychiatric, tumor diseases, etc.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction （one month after TAVR） | one month
  At 1-month follow-up, left ventricular ejection fraction was measured by echocardiography in patients with severe aortic stenosis complicated with heart failure after TAVR.

SECONDARY OUTCOMES:
Left ventricular size | one month
  At 1 month follow-up, the change of left ventricular size before and after TAVR.
left ventricular wall thickness | one month
  At 1 month follow-up, the change of left ventricular wall thickness before and after TAVR.
NT-proBNP | one month
  At 1 month follow-up, the change of NT-proBNP before and after TAVR.
Left ventricular global long axis strain | one month
  At 1 month follow-up, the change of left ventricular global long axis strain before and after TAVR.
aortic valve orifice area | one month
  At 1 month follow-up, the change of aortic valve orifice area before and after TAVR.
The result of 6-minute walking experiment | one month
  The result of 6-minute walking experiment was analyzed 1 month after TAVR.
Incidence of cardiovascular events | one month
  The incidence of cardiovascular disease was measured 1 month after TAVR.

CONTACTS AND LOCATIONS:
Overall Officials: guipeng an, M.D., Study Director — Qilu hospital of Shan Dong University
Locations (1):
- QIlu hospital of shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
We have no plans to share data

REFERENCES:
- [Result] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Result] Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart diseases: a population-based study. Lancet. 2006 Sep 16;368(9540):1005-11. doi: 10.1016/S0140-6736(06)69208-8. PMID 16980116
- [Result] Jorgensen K, Bech-Hanssen O, Houltz E, Ricksten SE. Effects of levosimendan on left ventricular relaxation and early filling at maintained preload and afterload conditions after aortic valve replacement for aortic stenosis. Circulation. 2008 Feb 26;117(8):1075-81. doi: 10.1161/CIRCULATIONAHA.107.722868. Epub 2008 Feb 11. PMID 18268152